CLINICAL TRIAL: NCT01098760
Title: A Phase IV, Single-arm, Open-label Study of Sorafenib (Nexavar®) in Advanced Hepatocellular Carcinoma (HCC)
Brief Title: Hepatocellular Carcinoma - Advanced Stage - Sorafenib Trial in Taiwanese Patients
Acronym: HATT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14898; HATT
Record Dates: First submitted 2010-04-01; First posted 2010-04-05 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Sorafenib; Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006) Sorafenib (Nexavar, BAY43-9006) + Nerison Fatty Ointment Sorafenib (Nexavar, BAY43-9006)+Neribas Fatty Ointment

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) Sorafenib (Nexavar, BAY43-9006) + Nerison Fatty Ointment Sorafenib (Nexavar, BAY43-9006)+Neribas Fatty Ointment — Orally taken Sorafenib tablets of 400mg (2x200mg) twice daily (bid) in a continuous schedule. - For patients in Nerisone subgroup: additionally prophylactic use of Nerisone Fatty Ointment (1 g of Nerisone contains 1 mg (0.1%) diflucortolone valerate) cream for hands and feet, twice daily for 3 weeks - For patients in Neribas subgroup: additionally prophylactic use of Neribas Fatty Ointment (non-corticosteroid containing) cream for hands and feet, twice daily for 3 weeks

SUMMARY:
This is a single-arm, open-label and post-authorization study to evaluate the safety and efficacy profile of sorafenib and to evaluate Child-Pugh status progression in subjects with advanced HCC treated with sorafenib in Taiwan.

In a subgroup of patients (hand-foot skin reaction (HFSR) study subgroup), this study also aims to test if topical corticosteroids as preventive counter-measure applied to hands and feet for the first 3 weeks during sorafenib treatment reduce incidence and severity of HFSR compared to a matching, corticosteroid-free cosmetic ointment, measured over the first 3 and 6 weeks of sorafenib treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented HCC (documentation of original biopsy for diagnosis is acceptable if tumor tissue is unavailable) or clinical diagnosis by American Association for the Study of Liver Disease (AASLD) criteria in cirrhotic patients is required. For subjects without cirrhosis, histological or cytological confirmation is mandatory.
* Unresectable advanced/or metastatic HCC not amenable to local treatment modalities
* Patients must have at least one tumor lesion that meets both of the following criteria:

  1. The lesion can be accurately measured in at least one dimension according to RECIST amendment (version 1.0)
  2. The lesion has not been previously treated with local therapy (such as surgery, radiation therapy, hepatic arterial therapy, chemoembolization, radiofrequency ablation, percutaneous ethanol injection, or cryoablation).
* Patients who have received local therapy such as surgery, radiation therapy, hepatic arterial embolization, chemoembolization, radiofrequency ablation, percutaneous ethanol injection, or cryoablation are eligible. Previously treated lesions will not be selected as target lesions. Local therapy must be completed at least 4 weeks prior to the baseline scan.
* Cirrhotic status of Child-Pugh Class A. Child-Pugh status should be calculated based on clinical findings and laboratory results during the screening period.
* Male or female patients >/= 18 years of age
* Patients who have a life expectancy of at least 12 weeks
* Patients who have an Eastern Cooperative Oncology Group (ECOG) performance score (PS) of 0,1 or 2
* Resolution of all acute toxic effects of any prior local treatment to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 grade </= 1
* The following laboratory parameters:

  1. Platelet count >/= 60 x 10^9/L
  2. Hemoglobin >/= 8.5 g/dL
  3. Total bilirubin </= 2.8 mg/dL
  4. Alanine transaminase (ALT) and aspartate aminotransferase (AST) </= 5 x upper limit of normal
  5. Serum creatinine </= 1.5 x the upper limit of normal
  6. Prothrombin time-international normalized ratio (INR) </=2.3 or PT </= 6 seconds above control.
* Patients who are being therapeutically anticoagulated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists. Close monitoring of at least weekly evaluations will be performed until INR is stable based on a measurement at pre dose, as defined by the local standard of care.

Exclusion Criteria:

* Previous or concurrent cancer that is distinct in primary site or histology from HCC, except cervical carcinoma in situ, treated basal cell carcinoma, or superficial bladder tumors (Ta, Tis &T1). Any cancer curatively treated > 3 years prior to entry is permitted.
* Renal failure requiring hemo- or peritoneal dialysis.
* History of cardiac disease:
* Congestive heart failure > New York Heart Association (NYHA) class 2
* Active coronary artery disease (myocardial infarction more than 6 months prior to study entry is permitted)
* Cardiac arrhythmias requiring anti-arrhythmic therapy other than β-blockers or digoxin)
* Uncontrolled hypertension, defined as systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg despite optimal medical management.
* Active, clinically serious infections (> grade 2 NCI-CTCAE, version 4.0), except HBV/HCV infections
* Known history of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)-related illness or serious acute or chronic illness
* Known central nervous system tumors, including metastatic brain disease
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry
* History of organ allograft
* Child-Pugh Class B or C
* Previous treatment with yttrium-90 spheres
* Clinically significant (ie, symptomatic) peripheral vascular disease
* Substance abuse or medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known or suspected allergy to the investigational agents or any agent given in association with this trial
* Patients unable to take oral medication, requiring intravenous alimentation, who have malabsorption syndrome or any other conditions affecting gastrointestinal absorption, or who have active peptic ulcer disease
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study
* Pregnant or breastfeeding patients. Women of childbearing potential must have a negative urine pregnancy test performed within 7 days prior to the start of study drug (assessed locally). Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial.
* Uncontrolled ascites (defined as not easily controlled with diuretic treatment)
* Patients with viral diseases (eg, varicella, herpes zoster); tuberculous or syphilitic processes in the areas to be treated; and hypersensitivity to the active substances or to any of the excipients will not be included into the HFSR study subgroup.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2010-08; Primary Completion 2013-03 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Time to progression | 30 months
Progression-free survival | 30 months
Overall survival | 30 months
Adverse event and serious adverse event (SAE) profiles | 30 months
Child-Pugh status progression | 30 months
Plasma Sorafenib exposure (AUC0-12) | 30 months
For subjects randomized into HFSR study subgroup: overall HFSR incidence in the first 3 weeks of Sorafenib treatment | 18 months

SECONDARY OUTCOMES:
For HFSR study subgroup: a mean HFSR grade determined at the end of the first 3 weeks of sorafenib treatment. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- Taiwan (6):
  - Chiayi City
  - Hualien County
  - Kaohsiung City
  - Taichung
  - Taipei
  - Taoyuan District